CLINICAL TRIAL: NCT03325933
Title: Resistance Training and Cardiometabolic Health
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19
Sponsor: Arizona State University (Other)
Responsible Party: Principal Investigator, Siddhartha Angadi, Assistant Professor, Arizona State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY00006617
Record Dates: First submitted 2017-10-13; First posted 2017-10-30 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Insulin Sensitivity; Endothelial Dysfunction; Blood Pressure
Keywords: insulin sensitivity; muscle; strength; resistance training; strength training; vascular function; arterial stiffness; glucose tolerance
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Resistance Training 1 (Experimental): Participants will perform resistance training with high training loads and low repetitions (high load/low rep resistance training).
  Interventions: Other: High Load/Low Rep Resistance Training
- Resistance Training 2 (Experimental): Participants will perform resistance training with low training loads and high repetitions (Low load/high rep resistance training).
  Interventions: Other: Low Load/High Rep Resistance Training
- Wait-list control (No Intervention): This group will be offered the option of participating in either experimental group after the study is completed.

INTERVENTIONS:
Other: High Load/Low Rep Resistance Training — Participants will be prescribed High Load/Low Rep resistance training.
  Arms: Resistance Training 1
Other: Low Load/High Rep Resistance Training — Participants will be prescribed Low Load/High Rep resistance training.
  Arms: Resistance Training 2

SUMMARY:
This study will investigate the relationship between resistance training load and repetitions on cardiometabolic outcomes. The primary objective of this clinical trial is to determine whether high load or low load resistance exercise training affects arterial stiffness in overweight or obese men and women. Our secondary objectives are to investigate the effects of high and low load RT on vascular function, cardiac structure, and markers of insulin sensitivity. Finally, we are going to preliminarily explore the effects of resistance training on intestinal bacteria.

DETAILED DESCRIPTION:
While it has been firmly established that aerobic exercise training is an effective modality for managing cardiometabolic disease risk, the influence of resistance training (RT) is not as well characterized. It is well established that RT improves muscular strength, size, cross sectional area, and bone mineral density. Alterations in muscle fiber type, glycolytic and oxidative enzyme profile, skeletal muscle proteins, and rates of protein synthesis also occur in response to RT and are obtained from skeletal muscle biopsies. Data from quasi-experimental studies suggest that moderate-to-high repetition RT with lower training loads may positively affect skeletal muscle proteins (Glucose Transporter Type 4 (GLUT4), Hexokinase 2 (HK2), and Adenylate kinase 2 (AK2) involved in insulin signaling in non-diabetic, obese men. However, data on high load, low rep RT on these variables is lacking. Thus, we will collect skeletal muscle biopsies to determine if changes in insulin signaling skeletal muscle proteins are present in response to both training with both high and low training loads. There is also a body of evidence suggesting that RT may improve VO2peak values in individuals with low baseline VO2peak values via a possible increase in capillary density, however, results are currently mixed. Low VO2peak values in overweight and obese individuals are positively associated with high risk of cardiovascular and all-cause mortality. Thus, we will measure VO2peak values to determine if (A) starting previously untrained obese individuals with RT can also improve VO2peak and (B) potential changes in VO2peak are load dependent. RT has also been reported to improve insulin sensitivity and central pressure. Additionally, aerobic exercise training may positively influence alterations in the intestinal microbiome, with no currently available evidence on the effects of RT, Although RT has been shown to be beneficial for improving arterial stiffness and insulin sensitivity, most of the available literature is based on protocols prescribing moderate-to-high repetitions and thus lower training loads. Thus, the effects of prescribing higher training loads on the aforementioned variables are not fully understood.

Increased arterial stiffness (as characterized by carotid-femoral pulse wave velocity (PWV) and augmentation index) is a clinical marker for cardiovascular disease and an independent risk factor for adverse cardiovascular events and all-cause mortality. Increased arterial stiffness has is positively associated with insulin resistance and type II diabetes. In the early stages of insulin resistance, peripheral insulin action, which occurs primarily in the skeletal muscle is impaired. This leads to a compensatory increase in insulin release in order to maintain glucose homeostasis, thus leading to hypertrophy of the pancreatic β cells. During the early stages of insulin resistance, fasting glucose levels will remain normal, with hyperglycemia manifesting in the later stages. Chronic hyperinsulinemia and hyperglycemia in turn cause increases in the renin-angiotensin aldosterone system as well expression of the angiotensin type I receptor in vascular tissue, thus stimulating VSMC proliferation, which leads to an increase in arterial stiffness. Chronic hyperglycemia and/or type II diabetes can lead to an increase in the production of advanced glycation end products (AGEs), which are proteins or lipids that become glycated due to exposure to glucose. Excessive production of AGEs can lead to an increase in collagen cross linking in the vascular walls, which thus leads to an increase in arterial stiffness.

Thus, it appears that increases in arterial stiffness occur due to perturbations in pulsatile shear and flow, which leads to abnormal turnover of scaffolding proteins, specifically excessive collagen production, and the proliferation of VSMCs, which results in a stiffer vasculature. This is exacerbated by the insulin resistant and/or hyperglycemic state due to an increase in local activity of the RAAS and expression of angiotensin I receptor activation in the vascular wall and an increase in age production, which leads to an increase in VSMCs and collagen cross-linking, respectively, thus further contributing to the development of a stiffer vasculature. These structural changes can have deleterious downstream consequences that include ischemic heart disease, myocardial infarction, and heart failure.

Current studies on the effects of RT on arterial stiffness have reported mixed results. It has been suggested that training with higher loads may cause greater increases in stiffness than training with lower loads due to greater acute elevations in blood pressure that occur with high load RT. Case control studies have reported that resistance trained young and middle aged non obese men demonstrated higher levels of arterial stiffness when compared to their aged-matched counterparts. Alternative cross-sectional studies reported that muscular strength was inversely related with arterial stiffness. Follow-up randomized control trials (RCT) investigated changes in arterial stiffness after several months of RT in non-obese, resistance training naïve adults. Improvements in central pressure, in the absence of changes in PWV, have been reported in non-diabetic obese adults after 12 weeks of RT but the study lacked an effective control group. Additionally, improvements in insulin sensitivity in non-diabetic obese males after 12 weeks of RT but was not a randomized controlled trial (RCT). Improvements in endothelial function has also been reported after six months of progressive RT that included both moderate and high training loads. This is significant because endothelial dysfunction is a downstream consequence of increased arterial stiffness, and thus an improvement in endothelial function, as measured by relative flow mediated dilation (%FMD), in response to RT is a reflects an improvement in vascular function, which is unlikely to occur in conjunction with an increase in vascular stiffness. To our knowledge, there are no current published RCTs on the effects of high load RT that have measured both arterial stiffness and endothelial function. This study will follow up on previous studies by comparing the effects of two distinct RT protocols (high load vs low load) on arterial stiffness as, measured by PWV and augmentation index, and endothelial function, as measured by %FMD, to a nonexercising control group.

A body of literature exists to suggest that morphological changes of the left ventricle take place in response to resistance training. Case control studies have reported that elite resistance trained athletes demonstrate evidence of left ventricular wall thickening. The increase in left ventricular wall thickness is referred to as concentric hypertrophy, which occurs in response to a chronic increase in afterload. This occurs in the presence of increased arterial stiffness, uncontrolled hypertension, and aortic stenosis, all of which can lead to heart failure (HF). RT induced concentric hypertrophy appears to be a physiological training adaptation, similar to the eccentric hypertrophy that takes place in response to aerobic training, and thus does not appear to be deleterious. Furthermore, current RCTs on the effects of RT on morphological changes of the LV suggest that this adaptation does not always occur or may occur in response to specific training volumes, frequencies, intensities, and/or over a longer training duration. Since the main outcome of this study is arterial stiffness, which is a precursor for concentric hypertrophy of the LV, we will also measure left ventricular wall thickness to see if A) morphological changes in the LV take place and B) if LV morphological changes are influenced by training load.

Thus, it appears that moderate training loads are shown to improve insulin sensitivity in obese individuals. This is significant because insulin resistance is a precursor to increases in arterial stiffness. However, the effects of training with higher loads on insulin sensitivity is a current gap in the literature. It has been previously proposed that high load RT may reduce arterial compliance and/or lead to concentric hypertrophy of the left ventricular walls. However, current evidence suggests that both moderate and high training loads improve endothelial function, without negatively affecting the left ventricular wall. Since endothelial dysfunction is a negative downstream consequence of an increase in arterial stiffness, it is unlikely that it would improve in conjunction with an increase in stiffness. Thus, this study will be the first to measure all of these variables to determine if and how they are influenced by training load.

The intestinal human microbiome is a recent target of interest due to its role in metabolic disease risk. Current evidence reports a link between cardiometabolic diseases and changes in the intestinal microbiota. The effects of exercise training on changes in the intestinal microbiome is also currently under investigation. Evidence in rat models currently suggest that voluntary and controlled aerobic exercise training is associated with favorable changes in the gut microbiome. However, human studies on the effects of exercise on the intestinal microbiome are currently lacking. .

The purpose of this study is to investigate the effects and potential differences between high load and low load RT on arterial stiffness. Based on the above described gaps in the literature the current study will serve as a follow up RCT to previous studies and will further explore the link between RT, arterial stiffness, and insulin sensitivity. From an exploratory stand-point we will examine changes if any in the gut microbiome following resistance training versus control. The proposed study will serve as a follow up RCT to investigate the differences between high load and low load RT on markers of arterial stiffness and insulin sensitivity. This study will also serve as the first RCT to investigate the long-term effects of RT in the intestinal microbiome. Studies investigating the effects of high load/low repetition RT on cardiometabolic biomarkers are currently lacking, with the current body of literature focusing on the effects of moderate and low loads and high repetitions, with limited data on the effects of high load RT.

ELIGIBILITY:
Inclusion Criteria:

* Male and female
* 18-55 years of age
* BMI 25-40
* No recent history of starting a structured exercise program or diet in the last 3 months

Exclusion Criteria:

* Current smoker and/or recreational drug user
* Answers "yes" to one or more questions on the Physical Activity Readiness Questionnaire
* Diagnosed diabetes, heart disease
* History of anabolic steroid use in the past six months
* Taking medications for treatment of diabetes, heart disease, and hypertension.
* Orthopedic or musculoskeletal contraindications to resistance training
* Unwilling to follow any aspect of the study protocol including blood sampling and weight training

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2017-09-21 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Arterial Stiffness | Change from Baseline Pulse Wave Velocity at 12 weeks
  Measured via pulse wave velocity

SECONDARY OUTCOMES:
Insulin Sensitivity | Change from Baseline Matsuda Index at 12 weeks
  Measured via oral glucose tolerance testing (OGTT)
Endothelial Function | Change from Baseline %FMD at 12 weeks
  Measured via flow mediated dilation (FMD)
Cardiac echocardiography | Changes in systolic and diastolic parameters from baseline to 12 weeks
  Measured using ultrasound
Isokinetic Strength | Change from Baseline isokinetic strength at 12 weeks
  Measured via dynamometry
Isometric Strength | Change from Baseline Isometric strength at 12 weeks
  Measured via dynamometry
Hexokinase | Change from Baseline in insulin signalling proteins at 12 weeks
  Measured via skeletal muscle biopsies
Insulin signaling proteins | Change from Baseline in insulin signaling proteins at 12 weeks
  Measured via skeletal muscle biopsies
Muscle Volume | Change from Baseline Muscle Volume at 12 weeks
  Measured via ultrasonography
Body Composition | Change from Baseline body composition at 12 weeks
  Measured via Dual X-Ray Absorptiometry (DXA)
Central Systolic Pressure | Change from Baseline Central Systolic Pressure at 12 weeks
  Measured via Pulse Wave Analysis
Central Diastolic Pressure | Change from Baseline Central Systolic Pressure at 12 weeks
  Measured via Pulse Wave Analysis

OTHER OUTCOMES:
Maximal Oxygen Consumption | Change from Baseline VO2peak at 12 weeks
  Measured via VO2peak testing using an integrated metabolic system.

CONTACTS AND LOCATIONS:
Overall Officials: Siddhartha S Angadi, PhD, Principal Investigator — Arizona State University
Locations (1):
- Arizona State University, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No
This data will be used primarily for a doctoral dissertation project as well as manuscript publication.

REFERENCES:
- [Background] Yang Q, Cogswell ME, Flanders WD, Hong Y, Zhang Z, Loustalot F, Gillespie C, Merritt R, Hu FB. Trends in cardiovascular health metrics and associations with all-cause and CVD mortality among US adults. JAMA. 2012 Mar 28;307(12):1273-83. doi: 10.1001/jama.2012.339. Epub 2012 Mar 16. PMID 22427615
- [Background] Safar ME, Czernichow S, Blacher J. Obesity, arterial stiffness, and cardiovascular risk. J Am Soc Nephrol. 2006 Apr;17(4 Suppl 2):S109-11. doi: 10.1681/ASN.2005121321. PMID 16565231
- [Background] Wildman RP, Mackey RH, Bostom A, Thompson T, Sutton-Tyrrell K. Measures of obesity are associated with vascular stiffness in young and older adults. Hypertension. 2003 Oct;42(4):468-73. doi: 10.1161/01.HYP.0000090360.78539.CD. Epub 2003 Sep 2. PMID 12953016
- [Background] Strasser B, Arvandi M, Pasha EP, Haley AP, Stanforth P, Tanaka H. Abdominal obesity is associated with arterial stiffness in middle-aged adults. Nutr Metab Cardiovasc Dis. 2015 May;25(5):495-502. doi: 10.1016/j.numecd.2015.01.002. Epub 2015 Jan 28. PMID 25770757
- [Background] Mitchell GF, Hwang SJ, Vasan RS, Larson MG, Pencina MJ, Hamburg NM, Vita JA, Levy D, Benjamin EJ. Arterial stiffness and cardiovascular events: the Framingham Heart Study. Circulation. 2010 Feb 2;121(4):505-11. doi: 10.1161/CIRCULATIONAHA.109.886655. Epub 2010 Jan 18. PMID 20083680
- [Background] Vlachopoulos C, Aznaouridis K, Stefanadis C. Prediction of cardiovascular events and all-cause mortality with arterial stiffness: a systematic review and meta-analysis. J Am Coll Cardiol. 2010 Mar 30;55(13):1318-27. doi: 10.1016/j.jacc.2009.10.061. PMID 20338492
- [Background] Ashor AW, Lara J, Siervo M, Celis-Morales C, Mathers JC. Effects of exercise modalities on arterial stiffness and wave reflection: a systematic review and meta-analysis of randomized controlled trials. PLoS One. 2014 Oct 15;9(10):e110034. doi: 10.1371/journal.pone.0110034. eCollection 2014. PMID 25333969
- [Background] Hellsten Y, Nyberg M. Cardiovascular Adaptations to Exercise Training. Compr Physiol. 2015 Dec 15;6(1):1-32. doi: 10.1002/cphy.c140080. PMID 26756625
- [Background] Miyachi M. Effects of resistance training on arterial stiffness: a meta-analysis. Br J Sports Med. 2013 Apr;47(6):393-6. doi: 10.1136/bjsports-2012-090488. Epub 2012 Jan 20. PMID 22267567
- [Background] Bertovic DA, Waddell TK, Gatzka CD, Cameron JD, Dart AM, Kingwell BA. Muscular strength training is associated with low arterial compliance and high pulse pressure. Hypertension. 1999 Jun;33(6):1385-91. doi: 10.1161/01.hyp.33.6.1385. PMID 10373221
- [Background] Miyachi M, Donato AJ, Yamamoto K, Takahashi K, Gates PE, Moreau KL, Tanaka H. Greater age-related reductions in central arterial compliance in resistance-trained men. Hypertension. 2003 Jan;41(1):130-5. doi: 10.1161/01.hyp.0000047649.62181.88. PMID 12511542
- [Background] Fahs CA, Heffernan KS, Ranadive S, Jae SY, Fernhall B. Muscular strength is inversely associated with aortic stiffness in young men. Med Sci Sports Exerc. 2010 Sep;42(9):1619-24. doi: 10.1249/MSS.0b013e3181d8d834. PMID 20195176
- [Background] Miyachi M, Kawano H, Sugawara J, Takahashi K, Hayashi K, Yamazaki K, Tabata I, Tanaka H. Unfavorable effects of resistance training on central arterial compliance: a randomized intervention study. Circulation. 2004 Nov 2;110(18):2858-63. doi: 10.1161/01.CIR.0000146380.08401.99. Epub 2004 Oct 18. PMID 15492301
- [Background] Rakobowchuk M, McGowan CL, de Groot PC, Bruinsma D, Hartman JW, Phillips SM, MacDonald MJ. Effect of whole body resistance training on arterial compliance in young men. Exp Physiol. 2005 Jul;90(4):645-51. doi: 10.1113/expphysiol.2004.029504. Epub 2005 Apr 22. PMID 15849230
- [Background] Yoshizawa M, Maeda S, Miyaki A, Misono M, Saito Y, Tanabe K, Kuno S, Ajisaka R. Effect of 12 weeks of moderate-intensity resistance training on arterial stiffness: a randomised controlled trial in women aged 32-59 years. Br J Sports Med. 2009 Aug;43(8):615-8. doi: 10.1136/bjsm.2008.052126. Epub 2008 Oct 16. PMID 18927168
- [Background] Okamoto T, Masuhara M, Ikuta K. Upper but not lower limb resistance training increases arterial stiffness in humans. Eur J Appl Physiol. 2009 Sep;107(2):127-34. doi: 10.1007/s00421-009-1110-x. Epub 2009 Jun 17. PMID 19533164
- [Background] Okamoto T, Masuhara M, Ikuta K. Effects of muscle contraction timing during resistance training on vascular function. J Hum Hypertens. 2009 Jul;23(7):470-8. doi: 10.1038/jhh.2008.152. Epub 2008 Dec 18. PMID 19092847
- [Background] Kawano H, Tanimoto M, Yamamoto K, Sanada K, Gando Y, Tabata I, Higuchi M, Miyachi M. Resistance training in men is associated with increased arterial stiffness and blood pressure but does not adversely affect endothelial function as measured by arterial reactivity to the cold pressor test. Exp Physiol. 2008 Feb;93(2):296-302. doi: 10.1113/expphysiol.2007.039867. Epub 2007 Oct 2. PMID 17911355
- [Background] Spence AL, Naylor LH, Carter HH, Buck CL, Dembo L, Murray CP, Watson P, Oxborough D, George KP, Green DJ. A prospective randomised longitudinal MRI study of left ventricular adaptation to endurance and resistance exercise training in humans. J Physiol. 2011 Nov 15;589(Pt 22):5443-52. doi: 10.1113/jphysiol.2011.217125. Epub 2011 Oct 3. PMID 21969450
- [Background] Cohen ND, Dunstan DW, Robinson C, Vulikh E, Zimmet PZ, Shaw JE. Improved endothelial function following a 14-month resistance exercise training program in adults with type 2 diabetes. Diabetes Res Clin Pract. 2008 Mar;79(3):405-11. doi: 10.1016/j.diabres.2007.09.020. Epub 2007 Nov 19. PMID 18006170
- [Background] Okamoto T, Masuhara M, Ikuta K. Effect of low-intensity resistance training on arterial function. Eur J Appl Physiol. 2011 May;111(5):743-8. doi: 10.1007/s00421-010-1702-5. Epub 2010 Oct 24. PMID 20972878
- [Background] Corretti MC, Anderson TJ, Benjamin EJ, Celermajer D, Charbonneau F, Creager MA, Deanfield J, Drexler H, Gerhard-Herman M, Herrington D, Vallance P, Vita J, Vogel R; International Brachial Artery Reactivity Task Force. Guidelines for the ultrasound assessment of endothelial-dependent flow-mediated vasodilation of the brachial artery: a report of the International Brachial Artery Reactivity Task Force. J Am Coll Cardiol. 2002 Jan 16;39(2):257-65. doi: 10.1016/s0735-1097(01)01746-6. PMID 11788217
- [Background] Tinken TM, Thijssen DH, Black MA, Cable NT, Green DJ. Time course of change in vasodilator function and capacity in response to exercise training in humans. J Physiol. 2008 Oct 15;586(20):5003-12. doi: 10.1113/jphysiol.2008.158014. Epub 2008 Aug 28. PMID 18755749
- [Background] Angadi SS, Mookadam F, Lee CD, Tucker WJ, Haykowsky MJ, Gaesser GA. High-intensity interval training vs. moderate-intensity continuous exercise training in heart failure with preserved ejection fraction: a pilot study. J Appl Physiol (1985). 2015 Sep 15;119(6):753-8. doi: 10.1152/japplphysiol.00518.2014. Epub 2014 Sep 4. PMID 25190739
- [Background] Croymans DM, Krell SL, Oh CS, Katiraie M, Lam CY, Harris RA, Roberts CK. Effects of resistance training on central blood pressure in obese young men. J Hum Hypertens. 2014 Mar;28(3):157-64. doi: 10.1038/jhh.2013.81. Epub 2013 Sep 5. PMID 24005959
- [Background] Cortez-Cooper MY, Anton MM, Devan AE, Neidre DB, Cook JN, Tanaka H. The effects of strength training on central arterial compliance in middle-aged and older adults. Eur J Cardiovasc Prev Rehabil. 2008 Apr;15(2):149-55. doi: 10.1097/HJR.0b013e3282f02fe2. PMID 18391640
- [Background] Julia M, Dupeyron A, Laffont I, Parisaux JM, Lemoine F, Bousquet PJ, Herisson C. Reproducibility of isokinetic peak torque assessments of the hip flexor and extensor muscles. Ann Phys Rehabil Med. 2010 Jun;53(5):293-305. doi: 10.1016/j.rehab.2010.05.002. Epub 2010 Jun 22. English, French. PMID 20634166
- [Background] Nagueh SF, Smiseth OA, Appleton CP, Byrd BF 3rd, Dokainish H, Edvardsen T, Flachskampf FA, Gillebert TC, Klein AL, Lancellotti P, Marino P, Oh JK, Alexandru Popescu B, Waggoner AD; Houston, Texas; Oslo, Norway; Phoenix, Arizona; Nashville, Tennessee; Hamilton, Ontario, Canada; Uppsala, Sweden; Ghent and Liege, Belgium; Cleveland, Ohio; Novara, Italy; Rochester, Minnesota; Bucharest, Romania; and St. Louis, Missouri. Recommendations for the Evaluation of Left Ventricular Diastolic Function by Echocardiography: An Update from the American Society of Echocardiography and the European Association of Cardiovascular Imaging. Eur Heart J Cardiovasc Imaging. 2016 Dec;17(12):1321-1360. doi: 10.1093/ehjci/jew082. Epub 2016 Jul 15. No abstract available. PMID 27422899
- [Background] Davis CC, Ellis TJ, Amesur AK, Hewett TE, Di Stasi S. IMPROVEMENTS IN KNEE EXTENSION STRENGTH ARE ASSOCIATED WITH IMPROVEMENTS IN SELF-REPORTED HIP FUNCTION FOLLOWING ARTHROSCOPY FOR FEMOROACETABULAR IMPINGEMENT SYNDROME. Int J Sports Phys Ther. 2016 Dec;11(7):1065-1075. PMID 27999721
- [Background] Abdul-Ghani MA, DeFronzo RA. Pathophysiology of prediabetes. Curr Diab Rep. 2009 Jun;9(3):193-9. doi: 10.1007/s11892-009-0032-7. PMID 19490820
- [Background] Micklesfield LK, Goedecke JH, Punyanitya M, Wilson KE, Kelly TL. Dual-energy X-ray performs as well as clinical computed tomography for the measurement of visceral fat. Obesity (Silver Spring). 2012 May;20(5):1109-14. doi: 10.1038/oby.2011.367. Epub 2012 Jan 12. PMID 22240726
- [Background] O'Sullivan O, Cronin O, Clarke SF, Murphy EF, Molloy MG, Shanahan F, Cotter PD. Exercise and the microbiota. Gut Microbes. 2015;6(2):131-6. doi: 10.1080/19490976.2015.1011875. Epub 2015 Mar 24. PMID 25800089
- [Background] Clarke SF, Murphy EF, O'Sullivan O, Lucey AJ, Humphreys M, Hogan A, Hayes P, O'Reilly M, Jeffery IB, Wood-Martin R, Kerins DM, Quigley E, Ross RP, O'Toole PW, Molloy MG, Falvey E, Shanahan F, Cotter PD. Exercise and associated dietary extremes impact on gut microbial diversity. Gut. 2014 Dec;63(12):1913-20. doi: 10.1136/gutjnl-2013-306541. Epub 2014 Jun 9. PMID 25021423
- [Background] Croymans DM, Paparisto E, Lee MM, Brandt N, Le BK, Lohan D, Lee CC, Roberts CK. Resistance training improves indices of muscle insulin sensitivity and beta-cell function in overweight/obese, sedentary young men. J Appl Physiol (1985). 2013 Nov 1;115(9):1245-53. doi: 10.1152/japplphysiol.00485.2013. Epub 2013 Aug 22. PMID 23970530
- [Background] Schram MT, Henry RM, van Dijk RA, Kostense PJ, Dekker JM, Nijpels G, Heine RJ, Bouter LM, Westerhof N, Stehouwer CD. Increased central artery stiffness in impaired glucose metabolism and type 2 diabetes: the Hoorn Study. Hypertension. 2004 Feb;43(2):176-81. doi: 10.1161/01.HYP.0000111829.46090.92. Epub 2003 Dec 29. PMID 14698999
- [Background] Ohnishi H, Saitoh S, Takagi S, Ohata J, Isobe T, Kikuchi Y, Takeuchi H, Shimamoto K. Pulse wave velocity as an indicator of atherosclerosis in impaired fasting glucose: the Tanno and Sobetsu study. Diabetes Care. 2003 Feb;26(2):437-40. doi: 10.2337/diacare.26.2.437. PMID 12547876
- [Background] Fleck SJ, Kraemer WJ. Resistance Training: Physiological Responses and Adaptations (Part 2 of 4). Phys Sportsmed. 1988 Apr;16(4):108-24. doi: 10.1080/00913847.1988.11709485. PMID 27457172
- [Background] Dickinson JM, Volpi E, Rasmussen BB. Exercise and nutrition to target protein synthesis impairments in aging skeletal muscle. Exerc Sport Sci Rev. 2013 Oct;41(4):216-23. doi: 10.1097/JES.0b013e3182a4e699. PMID 23873131
- [Background] Spence AL, Carter HH, Naylor LH, Green DJ. A prospective randomized longitudinal study involving 6 months of endurance or resistance exercise. Conduit artery adaptation in humans. J Physiol. 2013 Mar 1;591(5):1265-75. doi: 10.1113/jphysiol.2012.247387. Epub 2012 Dec 17. PMID 23247114
- [Background] Mihl C, Dassen WR, Kuipers H. Cardiac remodelling: concentric versus eccentric hypertrophy in strength and endurance athletes. Neth Heart J. 2008 Apr;16(4):129-33. doi: 10.1007/BF03086131. PMID 18427637
- [Background] Gaesser GA, Tucker WJ, Jarrett CL, Angadi SS. Fitness versus Fatness: Which Influences Health and Mortality Risk the Most? Curr Sports Med Rep. 2015 Jul-Aug;14(4):327-32. doi: 10.1249/JSR.0000000000000170. PMID 26166058
- [Background] Reaven GM. Banting lecture 1988. Role of insulin resistance in human disease. Diabetes. 1988 Dec;37(12):1595-607. doi: 10.2337/diab.37.12.1595. PMID 3056758
- [Background] Zieman SJ, Melenovsky V, Kass DA. Mechanisms, pathophysiology, and therapy of arterial stiffness. Arterioscler Thromb Vasc Biol. 2005 May;25(5):932-43. doi: 10.1161/01.ATV.0000160548.78317.29. Epub 2005 Feb 24. PMID 15731494